CLINICAL TRIAL: NCT07032948
Title: Safety and Efficacy Study of the First Domestically Produced FireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter Therapy for Rapid Arrhythmia With Tissue Temperature Measurement Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai MicroPort EP MedTech
Record Dates: First submitted 2025-06-12; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Rapid Arrhythmia; Atrial Fibrillation (AF); Paroxysmal Supraventricular Tachycardia (PSVT)
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid Arrhythmia（Paroxysmal supraventricular tachycardia and Atrial Fibrillation） (Experimental)
  Interventions: Device: FireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter、EasyStars™ High Density Mapping Catheter、Columbus™ 3D EP Navigation System

INTERVENTIONS:
Device: FireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter、EasyStars™ High Density Mapping Catheter、Columbus™ 3D EP Navigation System — All patients were treated withFireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter、EasyStars™ High Density Mapping Catheter and Columbus™ 3D EP Navigation System for rapid arrhythmia.

SUMMARY:
This project aims to evaluate the safety, efficacy, and cost-effectiveness of using FireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter to treat rapid arrhythmias.

DETAILED DESCRIPTION:
This project will conduct a clinical demonstration application study involving 300 cases, with the aim of evaluating the safety, efficacy, and cost-effectiveness of using FireMagic™ PreciSense™ 3D Microelectrode Ablation Catheter to treat rapid arrhythmias.

ELIGIBILITY:
1. Inclusion Criteria

1. Patient age between 18 and 75 years old, male or non-pregnant female;
2. Confirmed diagnosis of supraventricular tachycardia or atrial fibrillation requiring catheter radiofrequency ablation surgery;
3. Signed informed consent form approved by the ethics committee;
4. Willingness to undergo follow-up and evaluation as required by the protocol.

2. Exclusion Criteria Include:

1. Exclusion criteria for atrial fibrillation patients:

   Patients should not participate in this study if any of the following conditions apply:
   * Left atrial size ≥50 mm, left ventricular ejection fraction ≤40%;
   * Left atrial thrombus;
   * History of atrial septal repair or atrial myxoma;
   * History of cerebrovascular disease within the past 3 months (including stroke or transient ischaemic attack);
   * Cardiovascular events within the past 3 months (including acute myocardial infarction, coronary artery intervention or bypass surgery, artificial valve replacement or repair, or atrial or ventricular incision);
   * Acute or severe systemic infection;
   * Severe liver or kidney disease;
   * Significant bleeding tendency or haematological disorders;
   * Patients with other conditions deemed inappropriate for participation in this trial by the investigators.
2. Exclusion criteria for patients with ventricular tachycardia and supraventricular tachycardia:

Patients should not participate in this study if any of the following conditions apply:

* Left atrial size ≥50 mm and left ventricular ejection fraction ≤40%;
* History of atrial septal defect repair or atrial myxoma;
* Patients with cerebrovascular disease within the past 3 months (including stroke or transient ischaemic attack);
* Patients with cardiovascular events within the past 3 months (including acute myocardial infarction, coronary artery intervention or bypass surgery, artificial valve replacement or repair, or atrial or ventricular incision);
* Patients with acute or severe systemic infection;
* Patients with severe liver or kidney disease;
* Patients with a significant tendency to bleed or haematological disorders;
* Patients with other conditions deemed by the investigator to be unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
major evaluation indicators--Efficacy indicators | On the day of the surgery
  Immediate success rate of the investigational device in treating rapid arrhythmias;
Major evaluation indicators--Monitoring methods | On the day of the surgery
  Radiofrequency ablation treatment of rapid arrhythmias (such as supraventricular tachycardia and atrial fibrillation) using the trial device, with immediate ablation success determined based on the operator's professional experience combined with real-time intracardiac electrocardiogram display, followed by statistical analysis;
Major evaluation indicators--Safety indicators：Perioperative study of the incidence of adverse events related to medical devices | perioperative period
  Statistics on the incidence of adverse events related to surgical instruments during the perioperative period

SECONDARY OUTCOMES:
Changes in the surface temperature of the ablated tissue | During surgery
  extract multiple surface temperature data through tissue temperature measurement catheter microelectrodes and perform statistical analysis;
Changes in ablation point impedance | During surgery
  evaluate secondary indicators of tissue temperature measurement catheters, observe the impedance display of the radiofrequency ablation device, and record whether the impedance decreases during ablation